CLINICAL TRIAL: NCT04621630
Title: A Randomised, Double-Blind, Placebo-Controlled Study of Single and Multiple Ascending Doses of PN-235 in Healthy Volunteers
Brief Title: Pharmacokinetics of PN-235 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Protagonist Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: PN-235-01
Record Dates: First submitted 2020-10-29; First posted 2020-11-09 (Actual); Last update posted 2022-02-18 (Actual); Status verified 2022-02

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Bulk Drugs

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Part 1 blinded, Part 2 blinded, Part 3 unblinded
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Single Dose (Experimental): Single dose administration
  Interventions: Drug: PN-235; Drug: Placebo
- Multiple Dose (Experimental): Multiple dose administration
  Interventions: Drug: PN-235; Drug: Placebo
- Solid Dose Comparison (Experimental): Solid dose administartion
  Interventions: Drug: PN-235

INTERVENTIONS:
Drug: PN-235 — Active Drug
  Other Names: Active Drug
Drug: Placebo — Matching Placebo
  Arms: Multiple Dose; Single Dose

SUMMARY:
This Phase 1 study is designed to determine the safety, tolerability and pharmacokinetics of PN-235 in healthy volunteers. The study will be conducted in three parts: Part 1 is a single ascending dose study, Part 2 is multiple ascending dose study, and Part 3 is a randomized, crossover solid dose comparison and effect of food study.

DETAILED DESCRIPTION:
Part 1: Approximately 40 subjects randomized into 5 cohorts to receive PN-235 or placebo as single doses.

Part 2: Approximately 50 subjects enrolled into 5 cohorts to receive PN-235 or placebo once daily for 10 days.

Part 3: Twelve subjects will receive single doses of PN-235 in a 4-way, randomized, crossover fashion.

In total, approximately 102 subjects will participate.

ELIGIBILITY:
Key Inclusion Criteria:

* Subjects must have BMI between 18 and 32
* Subjects must be non-smokers or social smokers
* Subjects must comply with contraception requirements
* Subjects must be willing to consume meals provided by the clinical center

Key Exclusion Criteria:

* Subject must not have history of clinically significant endocrine, neurological, cardiovascular, hematological, hepatic, immunological, renal, respiratory, gastrointestinal or genitourinary abnormalities or diseases within previous 10 years
* Subjects must not have history of surgical resection of the stomach, small or large intestine
* Subjects must not have fever or symptomatic viral or bacterial infection within 2 weeks of screening
* Subjects must not have corrected QT greater than 450 msec in males and 470 msec in females
* Subjects must not test positive for Hepatitis C or B at Screening
* Subjects must refrain from use of prescription and non-prescription drugs and herbal remedies prior to initial dose of study drug and throughout the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2020-11-12 (Actual); Primary Completion 2021-09-19 (Actual); Study Completion 2021-10-13 (Actual)

PRIMARY OUTCOMES:
Safety of PN-235 | 10 days
  Number and severity of Adverse Events

SECONDARY OUTCOMES:
Pharmacokinetics (PK) of PN-235 in plasma | 10 days
  Peak concentration (Cmax) of PN-235
Area Under the Concentration (AUC) of PN-235 | 10 days
  AUC over 24 hours on Day 10 for PN-235

CONTACTS AND LOCATIONS:
Locations (1):
- Nucleus Network Melbourne Clinic, Melbourne, Australia

REFERENCES:
- [Derived] Knight B, Tammara B, Modi NB, Dallas S, Mardirosian S, Wang J, Laenen A, Leclercq L, DiLoreto K, Adriaenssen L, Moss D, Polidori D, Chaudhuri SR, Park S, Sensenhauser C, Ndifor A, Sukumaran S, Baguet T, Shi Y, Patel S, Geist B, Fourie A, Patch R, Sun C, Barros SA, Somani S, Monshouwer M. Translational Pharmacokinetics of Icotrokinra, a Targeted Oral Peptide that Selectively Blocks Interleukin-23 Receptor and Inhibits Signaling. Dermatol Ther (Heidelb). 2025 Sep;15(9):2495-2520. doi: 10.1007/s13555-025-01454-7. Epub 2025 Jul 8. PMID 40629250